CLINICAL TRIAL: NCT04391439
Title: Increased Heart Rhythm in Response to High-dose Intravenous Methylprednisolone Pulse Therapy of Moderate-to-severe Graves' Orbitopathy
Brief Title: Heart Rhythm After Intravenous Methylprednisolone Administration
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Piotr Miskiewicz, Assistant Professor, Medical University of Warsaw
Other Study IDs: IVMPheartrate
Record Dates: First submitted 2020-05-05; First posted 2020-05-18 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Graves Disease; Graves Ophthalmopathy; Heart Rhythm Disorder; Hypertension; Blood Pressure; Heart Failure
MeSH Terms: conditions — Graves Disease; Graves Ophthalmopathy; Hypertension; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All assays were performed in sera obtained from venous blood samples and analysed immediately after blood sampling in The Endocrinology Research Laboratory in the hospital. All samples were centrifugated for plasma immediately after delivery (15 min; 1000 xg) and separated for both categories (EDTA and heparin) - 2 x 400 ul for test tubes with protease inhibitors and 4 x 500 ul with no additives. Then all assays were frozen immediately to -70°C.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- active, moderate-to-severe GO: Each participant received IVMP according to EUGOGO recommendations (cumulative dose of methylprednisolone 4.5 g, treatment duration 12 weeks in single weekly intravenous pulses, first 6 weeks 0.5g of IVMP, next 6 weeks 0.25g of IVMP).
  Interventions: Drug: Intravenous Methylprednisolone

INTERVENTIONS:
Drug: Intravenous Methylprednisolone

SUMMARY:
High doses of intravenous (iv.) glucocorticoids (GCs) are commonly used as a treatment for many autoimmune and inflammatory disorders. According to the European Group on Graves' Orbitopathy (EUGOGO) guidelines, intravenous methylprednisolone (IVMP) is an accepted first-line agent for active, moderate-to-severe and very severe Graves' orbitopathy (GO). This treatment is proven to be more efficient and safer than oral GCs. However, some patients may experience adverse cardiovascular effects during the administration of iv. GCs, which in rare cases may even be fatal. There are limited data, mostly obtained from case reports, reporting the occurrence of cardiac arrhythmias, acute myocardial infarction or heart failure. Increased heart rhythm (HR) has drawn attention of researchers as a possible adverse effect correlated with IVMP. During this study, investigators performed 72-hours of Holter ECG and ambulatory blood pressure monitoring (ABPM) to evaluate the impact of IVMP on patients with moderate-to-severe GO, concerning HR and blood pressure (BP) changes. In order to elucidate possible mechanism of observed changes, researchers investigated the level of potassium in serum and urine and catecholamines (epinephrine, norepinephrine) in serum. All patients were treated routinely according to EUGOGO recommendations with standard doses of methylprednisolone with standard recommended schedule. Inclusion criterion for the therapy was according to EUGOGO guidelines active, moderate-to-severe and active GO (12 pulses of IVMP 6x0.5g followed by 6x0.25g every week).

DETAILED DESCRIPTION:
The clinical status of patients was evaluated before each pulse, including blood pressure monitoring, glucose level monitoring and symptoms of infection. HR and BP was measured continuously for 3 consecutive days (the day before, the day of IVMP and the day after IVMP) during 1st, 6th and 12th IVMP pulse, using 24-hour Holter ECG and ABMP. Serum laboratory tests for potassium, epinephrine and norepinephrine were measured 3 times the day before and the day of first IVMP pulse and 1 time the second and sixth day after 1st IVMP. Additionally, urine samples for potassium were collected 5 times the day of first IVMP pulse and 1 time the second and sixth day after 1st IVMP.

ELIGIBILITY:
Inclusion Criteria:

* active, moderate-to-severe GO according to EUGOGO classification
* euthyroidism
* completion of 12 IVMP pulses.

Exclusion Criteria:

* cardiovascular morbidity (such as chronic heart failure and/or coronary heart disease)
* uncontrolled hypertension (defined as systolic blood pressure (SBP) more than 140 mmHg and/or diastolic blood pressure (DBP) more than 90 mmHg)
* contraindications to IVMP therapy
* previous GCs treatment in the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the clinic for routine treatment of active, moderate-to-severe GO
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
24-hour Holter ECG Monitoring - 1st pulse mean HR | 72 hours
  Analysis of changes in mean HR between day before and day of 1st pulse of IVMP, day of 1st IVMP and day after 1st IVMP, day before and day after 1st IVMP
24-hour Holter ECG Monitoring - 6th pulse mean HR | 72 hours
  Analysis of changes in mean HR between day before and day of 6th pulse of IVMP, day of 6th IVMP and day after 6th IVMP, day before and day after 6th IVMP
24-hour Holter ECG Monitoring - 12th mean HR | 72 hours
  Analysis of changes in mean HR between day before and day of 12th pulse of IVMP, day of 12th IVMP and day after 12th IVMP, day before and day after 12th IVMP

SECONDARY OUTCOMES:
Serum potassium levels Day 0 - Day 1 | 48 hours
  Change in value of potassium between day before and day of 1st pulse of IVMP
Serum epinephrine levels Day 0 - Day 1 | 48 hours
  Change in value of epinephrine between day before and day of 1st pulse of IVMP
Serum norepinephrine levels Day 0 - Day 1 | 48 hours
  Change in value of norepinephrine between day before and day of 1st pulse of IVMP
Urine potassium levels Day 0 | 24 hours
  Change in value of potassium during the day of 1st pulse of IVMP
72-hour ambulatory blood pressure monitoring (ABPM) - 1st pulse mean BP | 72 hours
  Analysis of changes in mean BP between day before and day of 1st pulse of IVMP, day of 1st IVMP and day after 1st IVMP, day before and day after 1st IVMP
72-hour ambulatory blood pressure monitoring (ABPM) - 6th pulse mean BP | 72 hours
  Analysis of changes in mean BP between day before and day of 6th pulse of IVMP, day of 6th IVMP and day after 6th IVMP, day before and day after 6th IVMP
72-hour ambulatory blood pressure monitoring (ABPM) - 12th pulse mean BP | 72 hours
  Analysis of changes in mean BP between day before and day of 12th pulse of IVMP, day of 12th IVMP and day after 12th IVMP, day before and day after 12th IVMP

OTHER OUTCOMES:
Serum potassium levels Day 0 - Day 7 | 7 days
  Change in value of potassium between day before and sixth day after 1st pulse of IVMP
Serum potassium levels Day 0 - Day 2 | 72 hours
  Change in value of potassium between day of 1st IVMP and day after 1st IVMP, day before and day after 1st IVMP
Serum epinephrine levels Day 0 - Day 7 | 7 days
  Change in value of epinephrine between day before and sixth day after 1st pulse of IVMP
Serum epinephrine levels Day 0 - Day 2 | 72 hours
  Change in value of epinephrine between day of 1st IVMP and day after 1st IVMP, day before and day after 1st IVMP
Serum norepinephrine levels Day 0 - Day 7 | 7 days
  Change in value of epinephrine between day before and sixth day after 1st pulse of IVMP
Serum norepinephrine levels Day 0 - Day 2 | 72 hours
  Change in value of norepinephrine between day of 1st IVMP and day after 1st IVMP, day before and day after 1st IVMP
Urine potassium levels Day 1- Day 2 | 48 hours
  Change in value of epinephrine between day of 1st IVMP and day after 1st pulse of IVMP
Urine potassium levels Day 3 - Day 7 | 5 days
  Change in value of epinephrine between second and sixth day after 1st IVMP

IPD SHARING:
Plan to Share IPD: Yes
The collected data will be shared in a publication. It includes all laboratory results from all points of evaluation, results of 72-hour Holter ECG and 72-hour ABPM.
Time Frame: The results of the study will be published in 2020